CLINICAL TRIAL: NCT07397364
Title: Impact of Nurses' Behavior Change and Evidence-Based Practice Implementation on Quality Indicators in Intensive Care Units in Low- and Middle-Income Countries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Elhabashy, assistant professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-CU-EBP; 24K02733 (Other Grant/Funding Number: JSPS Scientific Research Grant)
Record Dates: First submitted 2026-01-21; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Ventilator-Associated Pneumonia (VAP); Central Line-Associated Bloodstream Infection; Pressure Ulcers (Hospital-acquired Pressure Injuries); Prolonged Intensive Care Unit Length of Stay; ICU Mortality (Survival Rate)
Keywords: Evidence-Based Practice; Nurses' Behavior Change; Intensive Care Unit; Quality Indicators; Ventilator-Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Development of the EBP educational program and materials:
  * The EBP education program (prototype, Table 1) is developed by this research team based on pedagogical method based on our research studies. Since nurses have not studied EBP and low motivation to change, this program introduces global comparison of quality indicators and online showing and exchange ICU-HUH situation by visual stimulation (awareness development).
  * After learning theories of EBP, each skill will be practiced in simulation training using manikins (Kyoto Kagaku, Japan & ICU-HUH originally developed materials). Using demonstration and redomnistration.
  * Skills training content will be provided from ICU- HUH (CN, Okamoto). Development of the in-ward training system will be also supported by nursing department of HUH under the framework of collaboration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Evidence-Based Practice Implementation) (Experimental): Participants in this arm will receive a structured evidence-based practice (EBP) education and behavior change program. The intervention includes theoretical training on EBP principles, simulation-based skills training, and supervised implementation of evidence-based ICU care bundles guided by the Plan-Do-Check-Act (PDCA) cycle. The program aims to improve nurses' competency, motivation, and adherence to evidence-based practices to reduce ICU-acquired complications.
  Interventions: Procedure: Evidence based practices bundles of care
- Control Group (Usual ICU Care) (No Intervention): Participants in this arm will continue providing routine ICU nursing care according to existing hospital policies and standard clinical guidelines. No additional EBP education or behavior change intervention will be provided during the study period. After completion of the study, participants in this arm will be offered the EBP education program.

INTERVENTIONS:
Procedure: Evidence based practices bundles of care — Participants in this arm will receive a structured evidence-based practice (EBP) education and behavior change program. The intervention includes theoretical training on EBP principles, simulation-based skills training, and supervised implementation of evidence-based ICU care bundles guided by the Plan-Do-Check-Act (PDCA) cycle. The program aims to improve nurses' competency, motivation, and adherence to evidence-based practices to reduce ICU-acquired complications.
  Arms: Intervention Group (Evidence-Based Practice Implementation)

SUMMARY:
Study title:

Impact of nurses' behavior change and implementing evidence-based practice to improve quality indicators in intensive care units in low-and middle-income countries

Background and Rationale:

Quality care is crucial for preventing adverse events and improving patient survival rates in healthcare settings, especially in the intensive care units (ICU). To improve patient outcomes, complying with evidence-based practice (EBP) and continuous monitoring of quality indicators by Plan-Do-Check- Act (PDCA) cycle is effective; in which "P: decide and plan target actions", "D: implement the plans", "C: measure and evaluate the indicators", and "A: discuss the next step for improvement". Regarding quality indicators at ICU, Japan has achieved the highest global survival rate with the fewest adverse events.

In a scoping review, when EBPs were implemented, 90% of the studies showed improved patient outcomes, and 94% found a positive return on investment. In ICU, EBP is essential for providing high-quality care, reducing errors, educating healthcare professionals, ensuring the efficacy of treatments, and fostering trust and good patient care relationships.

In Egypt, as a one of the low-and middle-income countries (LMICs), 59.9% of ICU patients had poor outcomes, with a 14.9% mortality rate. The incidence rate of total device- associated infections was 35.3/1000 device-days. The incidence of VAP is 38.4%, and it has reached 75% in some Egyptian hospitals; contrarily, in Japan, where Bundle care (evidence-based guideline) is strictly followed by nurses, the incidence of VAP is only 5.7%. EBP is hindered in LMICs by a lack of research infrastructure, a knowledge gap, poor nursing management, and limitation of resources. However, promoting this change will require increased advocacy of nurses, technical advancements, and integration into curricula and continuing education programs. Moreover, global collaboration is imperative for comprehensive development.

Objectives:

Primary Objective: Improve the quality of care in the ICU through implementation of EBP (indicated by selected quality indicators which assessed as routine work monthly in the selected ICU).

Secondary Objective: To enhance ICU nurses' professional competency in applying EBP.

The level of compatibility between the research proposal and the department's research goals.

There is a high level of compatibility between the research proposal and the department's research goals, particularly in terms of enhancing the competency of ICU staff through targeted training, improving the quality of care, and ultimately contributing to better patient outcomes.

The level of compatibility between the research proposal and the NCI 's research Plan.

The research proposal demonstrates a high level of compatibility with the NCI's research plan through the implementation of the latest evidence-based practices (EBP), standardized care protocols, and up-to-date clinical guidelines. It also aims to reduce contributing factors associated with increased morbidity and complication rates, thereby aligning with the institute's goals to advance patient safety and care quality.

- Study Design: An open- label, prospective, parallel-group (1:1), non-randomized controlled trial, with a pre- and post-design.

DETAILED DESCRIPTION:
National Cancer Institute - Cairo University Research Protocol

1. Proposed Study title: Impact of nurses' behavior change and implementing evidence-based practice to improve quality indicators in intensive care units in low-and middle-income countries 2. Principal investigator Name: Dr. Ahmed Shaban Mohammed 3. Date of application: June 29, 2025

1. Occupation Lecturer at Anesthesia and ICU and pain medicine National Cancer Institute
2. Emailing address : Dr.ahmed.shaban@gmail.com
3. Phone Number: 01222332541
4. Signature:

   5. Co-investigators Contact Information: Investigator (2) Professor Dr. Michiko Moriyama
   * Department Name: Graduate School of Biomedical and Health Sciences.
   * Faculty/ University: Hiroshima University, Japan
   * Phone Number: TEL +81-82-257-5365
   * Email Address: morimich@hiroshima-u.ac.jp
   * Signature:

   Investigator (3): Dr. Sameh Elsayed Elhabashy • Department Name: Lecturer at Nursing Education Department

   • Faculty/ University: Faculty of nursing, Cairo University

   • Phone Number: 01007653998
   * Email Address: Sameh17@cu.edu.eg Investigator (4): Professor Dr. Ekramy Mansour
   * Department Name: Professor of anesthesia and ICU and pain medicine Head of ICU unit
   * Faculty/ University: National Cancer Institute
   * Phone Number: +20 122 464 2810
   * Email Address: ekrameymansoure@yahoo.com

     5- Background and Rationale: Quality care is crucial for preventing adverse events and improving patient survival rates in healthcare settings, especially in the intensive care units (ICU). To improve patient outcomes, complying with evidence-based practice (EBP) and continuous monitoring of quality indicators by Plan-Do-Check- Act (PDCA) cycle is effective; in which "P: decide and plan target actions", "D: implement the plans", "C: measure and evaluate the indicators", and "A: discuss the next step for improvement". Regarding quality indicators at ICU, Japan has achieved the highest global survival rate with the fewest adverse events.

   In a scoping review, when EBPs were implemented, 90% of the studies showed improved patient outcomes, and 94% found a positive return on investment. In ICU, EBP is essential for providing high-quality care, reducing errors, educating healthcare professionals, ensuring the efficacy of treatments, and fostering trust and good patient care relationships.

   In Egypt, as a one of the low-and middle-income countries (LMICs), 59.9% of ICU patients had poor outcomes, with a 14.9% mortality rate. The incidence rate of total device- associated infections was 35.3/1000 device-days. The incidence of VAP is 38.4%, and it has reached 75% in some Egyptian hospitals; contrarily, in Japan, where Bundle care (evidence-based guideline) is strictly followed by nurses, the incidence of VAP is only 5.7%. EBP is hindered in LMICs by a lack of research infrastructure, a knowledge gap, poor nursing management, and limitation of resources. However, promoting this change will require increased advocacy of nurses, technical advancements, and integration into curricula and continuing education programs. Moreover, global collaboration is imperative for comprehensive development.

   6- Objectives: Primary Objective: Improve the quality of care in the ICU through implementation of EBP (indicated by selected quality indicators which assessed as routine work monthly in the selected ICU).

   Secondary Objective: To enhance ICU nurses' professional competency in applying EBP.

   7- The level of compatibility between the research proposal and the department's research goals.

   There is a high level of compatibility between the research proposal and the department's research goals, particularly in terms of enhancing the competency of ICU staff through targeted training, improving the quality of care, and ultimately contributing to better patient outcomes.

   The level of compatibility between the research proposal and the NCI 's research Plan.

   The research proposal demonstrates a high level of compatibility with the NCI's research plan through the implementation of the latest evidence-based practices (EBP), standardized care protocols, and up-to-date clinical guidelines. It also aims to reduce contributing factors associated with increased morbidity and complication rates, thereby aligning with the institute's goals to advance patient safety and care quality.

   8- Rationale of the study:

   • Critical role of ICU care: ICU patients are highly vulnerable; ensuring safe, evidence-based care is essential to reduce complications and improve survival.

   • Proven value of EBP: Global studies confirm that implementing Evidence-Based Practice (EBP) leads to better patient outcomes, fewer medical errors, and higher staff efficiency.

   • PDCA cycle effectiveness: The Plan-Do-Check-Act (PDCA) model supports continuous improvement in ICU settings, as successfully implemented in countries like Japan.

   • Egyptian ICU challenges:

   • Laking of nurse's awareness to the latest EBP and how to implement.

   • High rates of adverse outcomes as mentioned previously in the background.

   • Elevated rates of device-associated infections (e.g., ventilator-associated pneumonia).
   * Gap in EBP implementation: Barriers in LMICs like Egypt include limited resources, lack of EBP training, and absence of standardized guidelines.
   * Training as a solution: Empowering ICU nurses through targeted training in EBP can enhance their clinical competency, reduce infection rates, and improve overall care quality.

   Interventions (in details):

   Development of the EBP educational program and materials:

   ● The EBP education program (prototype, Table 1) is developed by this research team based on pedagogical method based on our research studies. Since nurses have not studied EBP and low motivation to change, this program introduces global comparison of quality indicators and online showing and exchange ICU-HUH situation by visual stimulation (awareness development).

   ●After learning theories of EBP, each skill will be practiced in simulation training using manikins (Kyoto Kagaku, Japan & ICU-HUH originally developed materials). Using demonstration and redomnistration.

   ●Skills training content will be provided from ICU- HUH (CN, Okamoto). Development of the in-ward training system will be also supported by nursing department of HUH under the framework of collaboration.

   Materials & Equipment for Simulation Training & Practice: For skill training at the sites, necessary materials and equipment will be prepared (currently, there is limited supply of the materials in study sites). For prevention of VAP, trachea tube with cuff, manometer, closed suction tube and oral care equipment would be prepared from Japan side (for teaching purpose). Then, the field hospitals will prepare them. Similarly, to prevent other adverse events, other equipment will be prepared from Japan side. the investigators educate and support the hospital for preparation (When economically difficult, alternative equipment would be created).

   11- Possible Risk and Adverse events: No significant risks or adverse events are anticipated for either patients or nurses as a result of this study.

   However, a minor risk may include: Increased time burden on nurses due to participation in training sessions which may temporarily affect their work schedule or routine tasks.

   To minimize this:

   • Training will be scheduled during non-peak hours whenever possible.

   • Nurse managers will be informed in advance to adjust duty rosters accordingly.

   • Continuous monitoring will be conducted to ensure that neither patient care nor staff well-being is compromised.

   14- Sample size estimation: For nurses: A total population sampling method will be used. All ICU nurses working in the selected ICU (approximately 35 nurses) who meet the inclusion criteria will be invited to participate in the intervention group. This approach ensures comprehensive representation and enhances the reliability of competency-related outcomes within the study setting.

   Sample size was estimated using G*Power software V.3.1.9.4 (Psychonomic Society, Madison, Wisconsin, USA), assuming α = 0.05, power (1-β err prob) = 0.75, and an effect size of 0.85. A sample size of 32 cases was required, divided into 16 patients as a control and 16 in study. with n1 = n2 = 42, after accounting for a 10% dropout or loss to follow-up rate. This sample size is deemed adequate based on a review of the literature.

   For patient: Given that no published studies comprehensively cover all the dependent variables collectively as assessed in our research, and to ensure a more accurate estimation of the required sample size for the patient group.

   15- Statistical analysis of data: Data will be expressed as mean and standard deviation (SD) for continuous variables and frequencies and percentages for categorical variables. The normality of data distribution was assessed using Shapiro-Wilk's test, histograms, and box plots. Baseline comparability between the control and intervention groups will be assessed using independent samples t-tests and chi-square tests. The incidence of VAP will be calculated as the number of new VAP cases per 1,000 ventilator days using the formula: (Number of new VAP cases / Total ventilator days) × 1000. A chi-square test will be used to compare the incidence between the pre- and post-intervention phases. An independent samples t-test will be employed to compare the difference between groups. Binary logistic regression analysis will be performed to evaluate the association between selected quality indicators and potential predictors, including group assignment (intervention or control). Statistical significance will be settled at a two-sided p-value of <0.05. All analyses were performed using SPSS version 27.0 (IBM, New York).

   16- Source of funding: The study will be self-funded

   17- Ethical committee approval:

   Protection of privacy and confidentiality:

   - The studies will be conducted according to the guidelines laid down in the Declaration of Helsinki and the Ethical Guidelines on Clinical Studies of the Ministry of Health.

   The proposed research studies will be initiated after its approval by the Institutional Review Boards (IRB) NCI. All trials will be registered in Clinical Trial registry.

   - Written consent will be obtained from nurses and patients who participate in the study, informing them of the purpose of the study, its methods, the voluntary nature of their participation, that they will not be disadvantaged if they do not consent, and that they may withdraw from the study during the course of the study.

   - Quality indicators are collected as one of the outcome measures of intervention studies. Therefore, approval from the IRBs to collect the data from the ICU database will also be obtained.

   - For the international benchmarking, approval of secondary use of the quality indicators will also be obtained from each IRB.
   * All the researchers including research assistants (RAs) who will directly involve in recruitment need to have Human Subject Protection Certificate (All researchers of PI, Co-I, R-Cos, and collaborating researchers from Cairo University, and Hiroshima University).

   the investigator shall assure that the privacy, anonymity, and confidentiality of data/information identifying the participant will be strictly maintained To avoid any disadvantage to patients due to not implementing the EBP, after each evaluation of one trial, the control group (nurses) will be educated on the EBP program.

ELIGIBILITY:
Inclusion Criteria:

For nurses:

* Willing to participate in this research.
* hold the existing position for at least three months.
* participants were required to have at least two years of critical care experience.

For patients:

- No specific inclusion criteria

Exclusion Criteria:

* for nurse:
* Nurses intending to leave their jobs within the study period (five months) were excluded.

For patients:

* admitted with Pressure ulcers.
* intubated outside the NCI
* Patients develop VAP in less than 48 hrs. after initiation of mechanical ventilation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ventilator-Associated Pneumonia (VAP) | Up to 5 months
  Incidence of ventilator-associated pneumonia measured as the number of new VAP cases per 1,000 ventilator-days in the ICU. using Ventilator-Associated Pneumonia (VAP) Assessment Sheet based on (CDC/NHSN) criteria
Incidence of Central Line-Associated Bloodstream Infection (CLABSI) | Up to 5 months
  Incidence of central line-associated bloodstream infection measured as the number of new CLABSI cases per 1,000 central line-days in the ICU. using Adult CLABSI Assessment & Audit Checklist. based on (CDC/NHSN) criteria

SECONDARY OUTCOMES:
Nurse Competency Score | Up to 5 months
  Nurses' competency in evidence-based practice and ICU care will be assessed using a validated competency assessment checklist. The total competency score will be calculated according to the checklist scoring system.
Incidence of Pressure Ulcers | Up to 5 months
  Incidence of hospital-acquired pressure ulcers measured as the number of new pressure ulcer cases among ICU patients during the study period. based on National Pressure Injury Advisory Panel (NPIAP).
Length of ICU Stay | Up to 5 months
  Length of stay in the intensive care unit measured in days from ICU admission to ICU discharge.
ICU Survival Rate | Up to 5 months
  Survival rate measured as the proportion of patients discharged alive from the ICU during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Michiko Moriyama, professor, Study Director — Hiroshima University
Locations (1):
- National Cancer Institute, Cairo, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No